CLINICAL TRIAL: NCT04408586
Title: Anti-Obesity Phentermine-Topiramate Extended Release Pharmacotherapy vs Placebo Among Patients Using a Wearable Activity Tracker.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Andres J. Acosta, M.D., Ph.D., Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19-011697
Record Dates: First submitted 2020-05-21; First posted 2020-05-29 (Actual); Results first posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Qsymia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phentermine - Topiramate Extended Release group (Active Comparator)
  Interventions: Drug: Phentermine-Topiramate Extended Release; Other: Online support system
- Placebo Group (Placebo Comparator)
  Interventions: Drug: Placebo; Other: Online support system

INTERVENTIONS:
Drug: Phentermine-Topiramate Extended Release — Dosing of 3.75/23 mg daily for 15 days, increased to 7.5/46 mg daily
  Other Names: Qsymia
  Arms: Phentermine - Topiramate Extended Release group
Drug: Placebo — Placebo looks exactly like the study drug, but it contains no active ingredient
  Arms: Placebo Group
Other: Online support system — VitalCare (VitalTech Affiliates LLC) is a digital health platform that allows remote collection of date from the wearable tracker and digital wellness devices used as part of this study. It also will allow subjects to document study medication compliance and will allow the remote visits to be conducted through a video conference between subjects and appropriate study team members.

SUMMARY:
Researchers are assessing the effects of weight loss medication vs a placebo among participants provided with a wearable activity tracker, digital wellness devices and lifestyle recommendations.

ELIGIBILITY:
Inclusion Criteria

* Adults with obesity (BMI >30Kg/m2); these will be otherwise healthy individuals with no unstable psychiatric disease and controlled comorbidities or other diseases.
* Age: 18-75 years.
* Gender: Men or women. Women of childbearing potential will have negative pregnancy tests within 48 hours of enrollment.
* Women of childbearing potential must agree to use a method of effective contraception during study participation.
* Subject must have an Apple iPhone 6s or later with iOS 13 or later and be willing to download the VitalCare (VitalTech Affiliates LLC) application from the Apple App Store.
* Able to provide written informed consent prior to any study procedures, and be willing and able to comply with study procedures

Exclusion Criteria

* History of Abdominal bariatric surgery
* Weight is greater than 450 lbs (204 kg)
* Recent use (within the last three months) of any antiobesity medication
* Recent weight change (gain or loss weight greater than 3% TBW in the last 3 months)
* Positive history of chronic gastrointestinal diseases, or systemic disease that could affect gastrointestinal motility, or use of medications that may alter gastrointestinal motility, appetite or absorption, e.g., orlistat, within the last 6 months.
* Significant untreated psychiatric dysfunction based upon screening with the Hospital Anxiety and Depression Inventory (HAD), and the Questionnaire on Eating and Weight Patterns (binge eating disorders and bulimia). If such a dysfunction is identified by an anxiety or depression score >11 or difficulties with substance or eating disorders, the participant will be excluded and given a referral letter to his/her primary care doctor for further appraisal and follow-up.
* Hypersensitivity or contraindication to the study medication.
* Participant unable or unwilling to follow protocol including use of the wearable activity tracker, digital wellness devices, VitalCare application, or unwilling to sign consent.
* Principal Investigator discretion

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-06-03 (Actual); Primary Completion 2022-06-13 (Actual); Study Completion 2022-10-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andres Acosta, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Campos A, Ghusn W, Cifuentes L, Sacoto D, Fansa S, Anazco D, Ricardo-Silgado ML, Hashem A, Schaefer M, Harmsen WS, Gunn HJ, Peterson C, Larsen D, Varghese ST, Hurtado MD, Acosta A. Addition of Phentermine-Topiramate to a Digitally Enhanced Lifestyle Intervention: A Double-Blind Randomized Clinical Trial. Obesity (Silver Spring). 2026 Jan 21. doi: 10.1002/oby.70108. Online ahead of print. PMID 41562388
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Phentermine - Topiramate Extended Release Group: Phentermine-Topiramate Extended Release: Dosing of 3.75/23 mg daily for 15 days, increased to 7.5/46 mg daily
  Online support system: VitalCare (VitalTech Affiliates LLC) is a digital health platform that allows remote collection of date from the wearable tracker and digital wellness devices that was used as part of this study. It also allowed subjects to document study medication compliance and allowed the remote visits to be conducted through a video conference between subjects and appropriate study team members.
- Placebo Group: Placebo: Placebo looks exactly like the study drug, but it contained no active ingredient
  Online support system: VitalCare (VitalTech Affiliates LLC) is a digital health platform that allows remote collection of date from the wearable tracker and digital wellness devices that was used as part of this study. It also allowed subjects to document study medication compliance and allowed the remote visits to be conducted through a video conference between subjects and appropriate study team members.
Period: Overall Study
Arm/Group | Phentermine - Topiramate Extended Release Group | Placebo Group
Started | 42 | 38
Completed | 42 | 38
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phentermine - Topiramate Extended Release Group | Placebo Group | Total
Number analyzed (Participants) | 42 | 38 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.4 (10.9) | 40.8 (10.2) | 42 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 32 | 68
  Male | 6 | 6 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 42 | 37 | 79
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 42 | 38 | 80

OUTCOME MEASURES:

1. Primary Outcome: Body Weight Change
Description: Change in weight calculated in kilograms.
Time Frame: baseline, 3 months
Measure: Mean (95% Confidence Interval); unit: kilograms
Arm/Group | Phentermine - Topiramate Extended Release Group | Placebo Group
Number analyzed (Participants) | 42 | 38
kilograms | -10.80 [-13.72 to -7.92] | -4.04 [-7.05 to -1.04]

2. Secondary Outcome: Body Weight Change
Description: Change in weight calculated in kilograms.
Time Frame: baseline, 12 months
Measure: Mean (95% Confidence Interval); unit: kilograms
Arm/Group | Phentermine - Topiramate Extended Release Group | Placebo Group
Number analyzed (Participants) | 42 | 38
kilograms | -15.32 [-18.65 to -12.00] | -5.85 [-9.40 to -2.30]

3. Secondary Outcome: Change in Step Count
Description: The change in the number of steps per day
Time Frame: baseline,12 months
Measure: Mean (95% Confidence Interval); unit: steps per day
Arm/Group | Phentermine - Topiramate Extended Release Group | Placebo Group
Number analyzed (Participants) | 42 | 38
steps per day | 1214 [-192 to 2620] | 2316 [807 to 3824]

4. Secondary Outcome: Change in Calories
Description: The change in calories burned per day
Time Frame: baseline, 12 months
Measure: Mean (95% Confidence Interval); unit: kcal per day
Arm/Group | Phentermine - Topiramate Extended Release Group | Placebo Group
Number analyzed (Participants) | 42 | 38
kcal per day | -193 [-356 to -30] | 60 [-127 to 247]

5. Secondary Outcome: Exercise Sessions
Description: The number of exercise sessions per week
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: sessions per week
Arm/Group | Phentermine - Topiramate Extended Release Group | Placebo Group
Number analyzed (Participants) | 42 | 38
sessions per week | 2.3 (1) | 2.1 (1)

6. Secondary Outcome: Tracker Usage
Description: The amount of time in minutes the tracker was used per week
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: minutes/week
Arm/Group | Phentermine - Topiramate Extended Release Group | Placebo Group
Number analyzed (Participants) | 42 | 38
minutes/week | 90 (15) | 94 (12)

7. Secondary Outcome: Change in SF-12 Physical Score (Health-related Quality Quality of Life)
Description: Quality of life SF12 physical score. The SF-12 is a well-validate measure of health-related quality of life; providing a physical and mental health component summary score. Min:0, Max: 100. Higher Score = Worse Outcome
Time Frame: baseline, 12 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Phentermine - Topiramate Extended Release Group | Placebo Group
Number analyzed (Participants) | 42 | 38
score on a scale | 1.99 [-0.34 to 4.32] | 0.57 [-1.76 to 2.90]

8. Secondary Outcome: Change in SF-12 Mental Score (Health-related Quality Quality of Life)
Description: Quality of life SF12 mental score. The SF-12 is a well-validate measure of health-related quality of life; providing a physical and mental health component summary score. Min:0, Max: 100. Higher Score = Worse Outcome.
Time Frame: baseline, 12 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Phentermine - Topiramate Extended Release Group | Placebo Group
Number analyzed (Participants) | 42 | 38
score on a scale | 0.42 [-1.66 to 2.50] | -1.48 [-3.56 to 0.60]

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from baseline to end of study, approximately 12 months for each subject
Arm/Group | Phentermine - Topiramate Extended Release Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/38
Other Adverse Events (participants affected / at risk) | 11/42 | 3/38
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phentermine - Topiramate Extended Release Group (N=42) | Placebo Group (N=38)
Paresthesia (Nervous system disorders) | 6 (6) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 3 (3) | 2 (2)
Dysgeusia (Nervous system disorders) | 3 (3) | 0 (0)
Insomnia (Psychiatric disorders) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-22): https://cdn.clinicaltrials.gov/large-docs/86/NCT04408586/Prot_SAP_000.pdf